CLINICAL TRIAL: NCT03286348
Title: Analysis of Nutrition During Chemoradiotherapy in Patients With Gastrointestinal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Hubei Cancer Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhen Zhang, MD, PHD, Fudan University
Other Study IDs: GINS-1001
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Nutritional Status; Gastrointestinal Cancer; Chemoradiotherapy
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the effectiveness of close and intense monitoring on nutritional status of gastrointestinal cancer patients during chemoradiotherapy (CRT), 500 CRT patients diagnosed with gastrointestinal system are going to be recruited into this prospective study. Patient-generated subjective global assessment (PG-SGA) scale and nutrition risk screening (NRS-2002) are used for nutritional assessment at the beginning and the end of CRT; Beside the nutritional parameters, Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) and gastric cancer module (QLQ-STO22) are used to measure quality of life in patients with gastric cancer while EORTC QLQ-C30 and Colorectal Cancer-Specific Quality of Life Questionnaire (QLQ-CR38) give assessment in colorectal cancer. The acute and late radiation toxicities were evaluated based on Conmon terminology criteria (CTC V3.0) and the toxicity criteria of RTOG/EORTC, respectively. Follow-ups every 3-6 months until three years after chemoradiotherapy are involved. Response Evaluation Criteria in Solid Tumors (RECIST) guidelines are used for response assessment. The primary endpoints are 3-year local control, disease-free survival, distant metastasis and overall survival rate.

ELIGIBILITY:
Inclusion Criteria for Gastric Cancer:

* pathological confirmed adenocarcinoma
* clinical stage T3-4 and/or N+ after radical surgery
* without distance metastases
* KPS >=70
* without previous radiotherapy
* sign the inform consent

Inclusion Criteria for Rectal Cancer:

* pathological confirmed adenocarcinoma
* clinical stage T3-4 and/or N+
* the distance from anal verge less than 12 cm
* without distance metastases
* KPS >=70
* without previous anti-cancer therapy
* sign the inform consent

Exclusion Criteria:

* pregnancy or breast-feeding women
* serious medical illness
* baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
* DPD deficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: gastric cancer patients and rectal cancer patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Local Control rate | From date of randomization until the date of first documented pelvic failure, assessed up to 3 years
  Number of participants with abdominal or pelvic failure after surgery, evaluated using Kaplan-Meier Curve

SECONDARY OUTCOMES:
Disease-free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhen Zhang, Shanghai, Shanghai Municipality, China